CLINICAL TRIAL: NCT00717626
Title: Pilot Study of Once-A-Day Prophylaxis for Youth and Young Adults With Severe Hemophilia A
Brief Title: Once-A-Day Prophylaxis for Youth and Young Adults With Severe Hemophilia A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000012140
Record Dates: First submitted 2008-07-14; First posted 2008-07-17 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Hemophilia A
Keywords: Hemophilia; Prophylaxis; Youth; Young Adults; Feasibility
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daily administration of low dose FVIII (Experimental): Low dose daily prophylaxis using FVIII products (e.g.Kogenate FS, Advate, or Humate-P, Recombinate, Helixate FS)
  Interventions: Drug: Kogenate FS, Advate, or Humate-P, Recombinate, Helixate FS

INTERVENTIONS:
Drug: Kogenate FS, Advate, or Humate-P, Recombinate, Helixate FS — Starting at the 4-month visit, subjects will receive 250 units per day (if their weight is < 50 kg.) or 500 units per day (weight ≥ 50 kg.) of their usual preparation of factor VIII.

SUMMARY:
The primary objective of this study is to test the feasibility of a large-scale clinical trial of once-daily prophylaxis. The secondary objectives are to collect clinical efficacy outcomes so that we can better plan a large-scale study; we will estimate the effect size and variability of effect and resource utilization of once-daily prophylaxis to allow us to set a sample size for a definitive trial.

DETAILED DESCRIPTION:
Hemophilia is an important and costly disorder; if left untreated, it may have serious consequences. The greatest impact of hemophilia occurs from recurrent bleeding into joints. The consequences of joint bleeding include pain associated with acute bleeding and later chronic arthropathy. Half of affected children with severe hemophilia have joint damage; joint damage is more frequent with increased bleeding. The prevention and treatment of bleeding is very expensive and therefore finding a cost-effective treatment is of high priority.

Worldwide, two major treatment strategies have been used to prevent arthropathy - on demand therapy and factor prophylaxis. The goal of prophylaxis is to convert the severe to the moderate phenotype by providing circulating factor activity of greater than 1%. Patients with greater than 1% circulating factor VIII activity rarely have spontaneous hemarthroses. Therefore, the goal of providing circulating factor at this level is to eliminate spontaneous hemarthroses. The term primary prophylaxis suggests using preventative factor VIII replacement from a very early age. The term secondary prophylaxis is used to describe the application of prophylaxis at a later disease stage. In this study, secondary prophylaxis will be used.

Once-daily prophylaxis is a novel application of hemophilia factor prophylaxis for youth and young adults. Before embarking on a costly definitive trial we feel that it is necessary to demonstrate that subjects will be willing to enroll and will be compliant with the therapy. Moreover, we need to establish an estimate of the effect of once-daily prophylaxis on bleeding rates, quality of life, and joint damage progression in order to design a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (<1% factor VIII)
* Age 12 to 24 years inclusive
* Male
* No current factor VIII inhibitor (an inhibitor will be defined as ≥ 0.6 Bethesda Units) within the past year
* Able to participate in a home infusion program with adequate peripheral venous access as assessed ny the treating investigator

Exclusion Criteria:

* Important co-morbidities (Acquired Immunodeficiency Syndrome or symptomatic HIV infection, symptomatic hepatitis B or C infection)
* Other concomitant acquired or congenital bleeding disorder (e.g. von Willebrand's Disease)
* Receiving factor VIII replacement through central venous catheter

Ages: 12 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feldman, MD,MSc,FRCPC, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Administration of Low Dose FVIII
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Region of Enrollment [Number; unit: participants]
  Canada | 14

OUTCOME MEASURES:

1. Primary Outcome: Hemophilia Joint Health Score (HJHS) 2.0
Description: Tool developed to assess joint health in persons with hemophilia (PWH) through several assessments of 9 items in the 6 index joints (elbows, knees, and ankles). It has been internationally validated and has demonstrated inter-observer and test-retest reliability supporting its use as an effective physical examination assessment tool for PWH.
  Range: 0 - 124 ( Best score = 0, Worst score = 124)
Time Frame: 4 months, 12 months
Population: Mean of differences between start of intervention (4 months) and end of study (12 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
score on a scale | 3.77 [0.63 to 6.91]

2. Primary Outcome: Functional Independence Score in Hemophilia (FISH)
Description: Tool for assessment of 8 areas of musculoskeletal (MSK) function in patients with hemophlia.
  Range: 0 - 32 ( Best score = 0, Worst score = 32)
Time Frame: 4 months, 12 months
Population: Mean of differences between start of intervention (4 months) and end of study (12 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
score on a scale | 0.31 [-0.41 to 1.02]

3. Primary Outcome: HRQoL Transformed Z-Score (Includes the Canadian Haemophilia Outcomes-Kids Life Assessment Tool (CHO-KLAT) and Haemo-QoL A)
Description: Canadian Haemophilia Outcomes-Kids Life Assessment Tool is a validated 35-item disease specific measure of Quality of Life in boys with hemophilia ages 4 - 17 yrs. Range: 0 - 100 ( Best score = 100, Worst score = 0)
  The Adult Haemo-QoL Questionnaire is a validated disease specific measure of Quality of Life in adults with hemophilia ages > 18 yrs. It is a 41-item questionnaire that considers how hemophilia affects 4 specific areas of their life. These areas include day-to-day activities, moods & feelings, work or school life, family life & social life, and hemophilia treatment. Range: 0 - 100 ( Best score = 0, Worst score = 100)
  The two measures were transformed into a Z-score to enable comparison across both HRQoL scores. A score of 0 represents no difference between the means, whereas a positive z-score would indicate an improvement in HRQoL between baseline and end of study.
Time Frame: 4 months, 12 months
Population: Mean of differences between start of intervention (4 months) and end of study (12 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
score on a scale | 0 [-0.64 to 0.64]

4. Primary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) . Version II
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) is an 11-item questionnaire used to evaluate patient satisfaction when starting a new medication and/or treatment. The areas of Effectiveness, Side-Effects, Convenience, and Global Satisfaction are assessed. A modified version (approved by developers) of the questionnaire with the deletion of side effects was used fro the purpose of the study.
  Effectiveness, Convenience, and Global Satisfaction all include the Range: 0 - 100 ( Best score = 0, Worst score = 100)
Time Frame: 4 months, 12 months
Population: Mean of differences between start of intervention (4 months) and end of study (12 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
score on a scale
  TSQM Effectiveness | -6.41 [-18.25 to 5.43]
  TSQM Convenience | -4.70 [-14.08 to 4.68]
  TSQM Global Satisfaction | -5.13 [-14.89 to 4.63]

5. Primary Outcome: The Previous Day Physical Activity Recall
Description: The Previous Day Physical Activity Recall is a well-validated assessment of habitual physical activity. Activity was reported on 1 weekend day, and 2 weekdays.The intensity of the activity was recorded in Metabolic Equivalents (METs) and categorized as Light (< 3.0 METs), Moderate (3.0 - 5.9 METs), Hard (6.0 - 8.9 METs), Very Hard (10.0 METs)
  Range: 0 - 10 METs per activity ( Best score = 10, Worst score = 0)
  MPA = Moderate Physical Activity VPA = Vigorous Physical Activity
Time Frame: 4 months and 12 months
Population: Mean of differences between start of intervention (4 months) and end of study (12 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
score on a scale
  Weekday 1 MPA | -0.15 [-2.24 to 1.94]
  Weekday 1 VPA | -0.69 [-3.65 to 2.26]
  Weekday 2 MPA | -0.15 [-2.54 to 2.24]
  Weekday 2 VPA | 0 [-5.1 to 5.1]
  Weekend MPA | -0.92 [-4.06 to 2.21]
  Weekend VPA | 2.31 [-1.76 to 6.38]

6. Secondary Outcome: Mean Yearly Factor Consumption of FVIII Product on Low Dose Daily Prophylaxis
Description: The mean yearly factor consumption of FVIII product on low dose daily prophylaxis was collected for comparison against standard prophylaxis (High dose alternate day treatment). Patient diaries indicating the amount of factor VIII product taken per daily infusion was collected on study.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: International Units (IU)
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
International Units (IU) | 211528 [176125.79 to 246930.61]

7. Primary Outcome: Total Number of Index Joint Bleeds
Description: The total number of index joint (elbows, knees, ankles) were extracted from the participant's (self-reported) diaries.
Time Frame: 4, 8, and 12 months
Measure: Median (Full Range); unit: Bleeds
Arm/Group | Daily Administration of Low Dose FVIII
Number analyzed (Participants) | 14
Bleeds
  4 months - Index joint bleeds | 0 [0 to 5]
  8 months - Index joint bleeds | 0 [0 to 5]
  12 months - Index joint bleeds | 0 [0 to 12]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a duration of 1 year.
Description: An adverse event log was maintained for each participant to identify and report any of the following:
  1. All-Cause Mortality
  2. Serious Adverse Events
  3. Other Adverse Events
Arm/Group | Daily Administration of Low Dose FVIII
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No